CLINICAL TRIAL: NCT02655601
Title: A Phase 2 Trial for Patients With Newly Diagnosed High Grade Glioma Treated With Concurrent Radiation Therapy, Temozolomide, and BMX-001
Brief Title: Trial of Newly Diagnosed High Grade Glioma Treated With Concurrent Radiation Therapy, Temozolomide and BMX-001
Acronym: BMX-HGG
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioMimetix JV, LLC (Industry)
Collaborators: Duke Cancer Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMX-HGG-001
Record Dates: First submitted 2016-01-12; First posted 2016-01-14 (Estimated); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: High Grade Glioma; Astrocytoma, Grade III; Glioblastoma
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma | interventions — Mn(III) meso-tetrakis(N-n-butoxyethylpyridinium-2-yl)porphyrin; Radiotherapy; Temozolomide

STUDY DESIGN:
Intervention Model Description: There is 1 arm of subjects enrolled in Phase 1 (all subjects receiving the study drug + SOC). In Phase 2, subjects are enrolled in two arms (Arm A: SOC + BMX-001 and Arm B: SOC alone)
Masking Description: Phase 1 - Single Arm Phase 2- Randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 2 Arm A: Radiation Therapy, TMZ and BMX-001 (Experimental): Patients will receive standard of care radiation therapy plus temozolomide (TMZ). BMX-001 will be given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks. A total of 80 subjects will receive BMX-001 in this phase.
  Interventions: Drug: BMX-001; Radiation: Radiation Therapy; Drug: Temozolomide
- Phase 2 Arm B: Radiation Therapy and TMZ (Active Comparator): In this arm, one-half of the study subjects will not receive BMX-001 but will undergo all components of standard therapy (radiation therapy plus temozolomide [TMZ]). A total of 80 subjects will be in this study arm.
  Interventions: Radiation: Radiation Therapy; Drug: Temozolomide
- Phase 1 (Experimental): All subjects enrolled will receive BMX-001 at one of 4 different dose levels. BMX-001 will be given by subcutaneous injection with a loading dose given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses (half the dosing dose) for a total of 8 weeks. Subjects will also undergo standard therapy (radiation therapy plus temozolomide [TMZ])
  Interventions: Drug: BMX-001; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Drug: BMX-001 — BMX-001 consists of a porphyrin ring with pyridyl groups attached at each of the four methane bridge carbons. The nitrogen in the pyridyl ring is at the 2 position and has a side chain consisting of six carbons with an ether linkage. A manganese atom is chelated into the porphyrin ring and is the active center of the molecule. This molecule is an enzymatic scavenger of free radical species operating at close to diffusion-limited rates.
  Other Names: manganese butoxyethyl pyridyl porphyrin
  Arms: Phase 1; Phase 2 Arm A: Radiation Therapy, TMZ and BMX-001
Radiation: Radiation Therapy — RT will be delivered in daily fractions of 1.8-2 Gy given 5 days a week for 6 weeks for a total of 59.4-60 Gy.
Drug: Temozolomide — Initially, temozolomide (TMZ) will be dosed at 75 mg/m2 orally daily for 42 days. Two weeks after the completion of chemoradiation, patients will transition to adjuvant chemotherapy with TMZ dosed at 150-200 mg/m2 orally for 5 days of a 28-day cycle for a total of 12 cycles.
  Other Names: TMZ

SUMMARY:
This is a Phase 2 study of newly diagnosed patients with high grade glioma (HGG) undergoing standard radiation therapy and temozolomide treatment. BMX-001 added to radiation therapy and temozolomide has the potential not only to benefit the survival of high grade glioma patients but also to protect against deterioration of cognition and impairment of quality of life. BMX-001 will be given subcutaneously first with a loading dose zero to four days prior to the start of chemoradiation and followed by twice a week doses at one-half of the loading dose for the duration of radiation therapy plus two weeks. Both safety and efficacy of BMX-001 will be evaluated. Impact on cognition will also be assessed. Eighty patients will be randomized to the treatment arm that will receive BMX-001 while undergoing chemoradiation and 80 patients randomized to receive chemoradiation alone. The sponsor hypothesizes that BMX-001 when added to standard radiation therapy and temozolomide will be safe at pharmacologically relevant doses in patients with newly diagnosed high grade glioma. The sponsor also hypothesizes that the addition of BMX-001 will positively impact the overall survival and improve objective measures of cognition in newly diagnosed high grade glioma patients.

DETAILED DESCRIPTION:
160 patients will be enrolled and randomized with a treatment arm allocation ratio of 1:1 in the Phase 2 study. At enrollment, patients will be assessed with medical history, physical/neurological examinations, standard laboratory evaluations (CBC with differential and comprehensive metabolic panel (CMP)), baseline brain MRI with and without gadolinium, cognitive testing and patient-reported outcome questionnaires of HRQoL. On the first day of BMX-001 (loading dose), patients will be evaluated with medical history, patient physical/neurological examinations, and standard laboratory evaluations (CBC with differential and CMP), and ECG. Patients in Arm A will be administered BMX-001 subcutaneously first as a loading dose before the start of chemoradiation and then at maintenance dose (50% of the loading dose) twice a week for 8 weeks. Because oxidative stress continues to occur for up to several weeks following RT, the proposed protocol includes administering BMX-001 both before the start of RT and continuing for 2 weeks after the completion of RT and TMZ. TMZ will be dosed at 75 mg/m2 orally daily for 42 days and RT will be delivered in daily fractions of 1.8-2 Gy given 5 days a week for 6 weeks for a total of 59.4-60 Gy. During standard RT and TMZ, CBC with differential and CMP will be obtained weekly. Two weeks after the completion of standard RT and TMZ and every 8 weeks during adjuvant TMZ, patients will be evaluated with the following: medical history, physical/neurological examinations, Brain MRI with and without gadolinium, cognitive testing and patient-reported outcome questionnaires of HRQoL. Two weeks after the completion of chemoradiation, patients will transition to adjuvant chemotherapy with TMZ dosed at 150-200 mg/m2 orally for 5 days of a 28-day cycle for a total of 12 cycles. In light of the findings that BMX-001 can spare radiation-induced hair loss in a mouse model [41], we will evaluate and describe hair loss as an exploratory outcome in HGG patients by evaluating hair at baseline and then every 8 weeks. Patients will be discontinued from the study if they experience progression of disease, death or withdraw informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed diagnosis of World Health Organization (WHO) grade III or IV malignant glioma
* Subjects must be planning to start standard of care radiation therapy and chemotherapy
* Subjects must be within 12 weeks of last major neurosurgical procedure for the high-grade glioma (craniotomy, open biopsy, or stereotactic biopsy)
* Subjects must have had a definitive resection with residual radiographic contrast enhancement on post-resection CT or MRI of less than or equal to 3 cm in any two perpendicular planes on any images
* Age * 18 years
* Karnofsky Performance Status (KPS) ≥ 70%
* Hemoglobin ≥ 9.0 g/dl, absolute neutrophil count (ANC) ≥ 1,500 cells/µl, platelets ≥ 125,000 cells/µl
* Serum creatinine ≤ 1.5 mg/dl, serum glutamate oxaloacetate transaminase (SGOT) and bilirubin ≤ 1.5 times upper limit of normal
* Signed informed consent approved by the Institutional Review Board
* If sexually active, patients must agree to use appropriate contraceptive measures for the duration of the study and for 12 months afterwards as stated in the informed consent
* Stable and/or decreasing dose of corticosteroids for greater than or equal to 7 days.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Active infection requiring IV antibiotics 7 days before enrollment
* Signs of wound-healing problems or infection at the craniotomy/biopsy site.
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
* Prior treatment with radiotherapy or chemotherapy for a brain tumor, irrespective of the grade of the tumor
* Evidence of > grade 1 CNS hemorrhage on baseline MRI on CT scan
* Systemic treatment with inducers or strong inhibitors of cytochrome P450 within four days before enrollment or planned treatment during the time period of the study.
* Metal in the body (except dental fillings) e.g., pacemaker, infusion pump, metal aneurysm clip, metal prosthesis, joint, rod or plate.
* Severe allergy to contrast agent.
* Inadequately controlled hypertension
* Active or history of postural hypotension and autonomic dysfunction
* Clinically significant (i.e. active) cardiovascular disease or cerebrovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
* History or evidence upon physical/neurological examination of central nervous system disease (e.g. seizures) unrelated to cancer unless adequately controlled by medication or potentially interfering with protocol treatment
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 milliseconds (ms) (CTCAE grade 1)
* A known history of additional risk factors for Torsades de Pointes (TdP) (e.g., congestive heart failure, hypokalemia, known family history of Long QT Syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2023-08-17 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Peters, MD, PhD, Principal Investigator — Duke Cancer Institute
Locations (9):
- United States (9):
  - University of Alabama- Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Kentucky, Lexington, Kentucky
  - St. Luke's Hospital, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke Cancer Institute, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones LW, Cohen RR, Mabe SK, West MJ, Desjardins A, Vredenburgh JJ, Friedman AH, Reardon DA, Waner E, Friedman HS. Assessment of physical functioning in recurrent glioma: preliminary comparison of performance status to functional capacity testing. J Neurooncol. 2009 Aug;94(1):79-85. doi: 10.1007/s11060-009-9803-x. Epub 2009 Feb 11. PMID 19212703
- [Background] Moulder JE, Cohen EP. Future strategies for mitigation and treatment of chronic radiation-induced normal tissue injury. Semin Radiat Oncol. 2007 Apr;17(2):141-8. doi: 10.1016/j.semradonc.2006.11.010. PMID 17395044
- [Derived] Gad SC, Sullivan DW Jr, Spasojevic I, Mujer CV, Spainhour CB, Crapo JD. Nonclinical Safety and Toxicokinetics of MnTnBuOE-2-PyP5+ (BMX-001). Int J Toxicol. 2016 Jul;35(4):438-53. doi: 10.1177/1091581816642766. Epub 2016 Apr 20. PMID 27098749

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 17 subjects were enrolled at 1 center for Phase 1. For Phase 2, 160 subjects were enrolled at 9 clinical centers in the US (mostly comprising university and top tier HGG treatment facilities.)
Pre-assignment Details: Phase 1 was a dose escalation study. Phase 1 participants did not participate in Phase 2.
  In Phase 2, patients were considered to have completed treatment in Arm A if they completed SOC chemoradiation and received the study drug, BMX-001 for at least 6 weeks, or 13 doses. In Arm B, patients were considered to have completed treatment if they completed SOC chemoradiation.
Groups:
- Phase 1 BMX-001 7 mg Loading Dose/3.5 mg Biw Dose: BMX-001 was administered subcutaneously as a loading dose before starting concurrent standard of care chemoradiation. After the loading dose, the dose levels were given two times per week for 8 weeks. The starting dose level was a 7 mg loading dose followed by 3.5 mg maintenance doses twice a week for up to 8 weeks.
- Phase 1 BMX-001 14 mg Loading Dose/7 mg Biw Dose: BMX-001 was administered subcutaneously as a loading dose before starting concurrent standard of care chemoradiation. After the loading dose, the dose levels were given two times per week for 8 weeks. The second dose level was a 14 mg loading dose followed by 7 mg maintenance doses twice a week for up to 8 weeks.
- Phase 1 BMX-001 28 mg Loading Dose/14 mg Biw Dose: BMX-001 was administered subcutaneously as a loading dose before starting concurrent standard of care chemoradiation. After the loading dose, the dose levels were given two times per week for 8 weeks. The third dose level was a 28 mg loading dose followed by 14 mg maintenance doses twice a week for up to 8 weeks.
- Phase 1 BMX-001 42 mg Loading Dose/20 mg Biw Dose: BMX-001 was administered subcutaneously as a loading dose before starting concurrent standard of care chemoradiation. After the loading dose, the dose levels were given two times per week for 8 weeks. The fourth dose level was a 42 mg loading dose followed by 20 mg maintenance doses twice a week for up to 8 weeks.
- Ph 2 Radiation Therapy, TMZ and BMX-001: Patients received standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks. A total of 80 subjects were eligible to receive BMX-001 in this phase.
- Ph 2 Radiation Therapy and TMZ: In this arm, one-half of the study subjects did not receive BMX-001 but underwent all components of standard therapy (radiation therapy plus temozolomide [TMZ]). A total of 80 subjects were eligible for inclusion in this study arm.
Period: Overall Study
Arm/Group | Phase 1 BMX-001 7 mg Loading Dose/3.5 mg Biw Dose | Phase 1 BMX-001 14 mg Loading Dose/7 mg Biw Dose | Phase 1 BMX-001 28 mg Loading Dose/14 mg Biw Dose | Phase 1 BMX-001 42 mg Loading Dose/20 mg Biw Dose | Ph 2 Radiation Therapy, TMZ and BMX-001 | Ph 2 Radiation Therapy and TMZ
Started | 4 | 3 | 6 | 4 | 80 | 80
Completed | 3 | 3 | 6 | 3 | 74 | 71
Not Completed | 1 | 0 | 0 | 1 | 6 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 8
Not completed — Treatment delayed too long per protocol due to adverse events | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled in the Phase 1 dose escalation study + the Phase 2 randomized study
Groups:
- Phase 1 Dose Level 1: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001: Dose escalation study. Patients received standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 7 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks.
- Phase 1 Dose Level 2: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001: Dose escalation study. Patients received standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 14 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks.
- Phase 1 Dose Level 3: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001: Dose escalation study. Patients received standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks.
- Phase 1 Dose Level 4: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001: Dose escalation study. Patients received standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of42 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks.
- Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001: Patients received standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks. A total of 80 subjects were eligible to receive BMX-001 in this phase.
- Arm B: Ph 2 Radiation Therapy and TMZ: In this arm, one-half of the study subjects did not receive BMX-001 but underwent all components of standard therapy (radiation therapy plus temozolomide [TMZ]). A total of 80 subjects were eligible for inclusion in this study arm.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001 | Phase 1 Dose Level 2: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001 | Phase 1 Dose Level 3: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001 | Phase 1 Dose Level 4: Radiation Therapy, TMZ and BMX-001, All Patients Received BMX-001 | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ | Total
Number analyzed (Participants) | 4 | 3 | 6 | 4 | 80 | 80 | 177
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.5 (13.1) | 61.3 (2.1) | 64.3 (8.8) | 50 (24.7) | 52.69 (13.55) | 54.39 (14.23) | 53.54 (13.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 1 | 35 | 25 | 68
  Male | 2 | 2 | 2 | 3 | 45 | 55 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 3 | 4
  Not Hispanic or Latino | 4 | 3 | 6 | 4 | 79 | 76 | 172
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 2 | 4
  White | 4 | 3 | 6 | 3 | 75 | 72 | 163
  More than one race | 0 | 0 | 0 | 0 | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 6 | 4 | 80 | 80 | 177
WHO 2021 Histology [Count of Participants; unit: Participants] — The World Health Org (WHO) 2021 grading criteria for brain tumors provide an updated, classification system that stratifies central nervous system (CNS) tumors. This classification refines previous grading methods (prior to years 2021) by incorporating molecular markers to improve diagnostic accuracy, prognostic prediction, and therapeutic decision-making. The key criteria include: Histopathology, Molecular Markers, IDH mutation status, and other mutations, alterations, and amplifications.
  Ph 1 subjects were enrolled prior to the 2021 revision in criteria, this is only valid for ph 2. Population: This measurement was not in existence for Phase 1 and is only applicable to Phase 2
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 80 | 80 | 160
    Glioblastoma, IDH-wildtype | 0 | 0 | 0 | 0 | 55 | 56 | 111
    Astrocytoma, IDH-mutant | 0 | 0 | 0 | 0 | 17 | 15 | 32
    Oligodendroglioma, IDH-mutant, and 1p/19q-codeleted | 0 | 0 | 0 | 0 | 4 | 6 | 10
    Glioblastoma, NOS | 0 | 0 | 0 | 0 | 2 | 1 | 3
    Glioblastoma, IDH-wildtype, gliosarcoma subtype | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Ganglioglioma | 0 | 0 | 0 | 0 | 0 | 1 | 1
    Glioblastoma, IDH-wildtype, giant cell subtype | 0 | 0 | 0 | 0 | 1 | 0 | 1
    Pleomorphic Xanthoastrocytoma | 0 | 0 | 0 | 0 | 1 | 0 | 1
WHO 2021 Tumor Grade [Count of Participants; unit: Participants] — WHO Grade 3: Includes anaplastic astrocytomas (IDH-mutant), anaplastic oligodendrogliomas (IDH-mutant, 1p/19q-codeleted).
  WHO Grade 4: Includes glioblastoma (IDH-wildtype), astrocytoma (IDH-mutant, grade 4), and diffuse midline glioma (H3 K27-altered).
  Ph 1 subjects were enrolled prior to the 2021 revision in criteria, this is only valid for ph 2 Population: This measurement for 2021 WHO grading was not applicable at the time of Phase 1, and only works for Phase 2
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 80 | 80 | 160
    Grade 4 | 0 | 0 | 0 | 0 | 65 | 67 | 132
    Grade 3 | 0 | 0 | 0 | 0 | 15 | 13 | 28
WHO 2016 Histology [Count of Participants; unit: Participants]
  Glioblastoma Multiforme | 3 | 3 | 6 | 4 | 61 | 64 | 141
  Anaplastic astrocytoma | 0 | 0 | 0 | 0 | 11 | 7 | 18
  Anaplastic oligodendroglioma | 0 | 0 | 0 | 0 | 4 | 6 | 10
  Giant Cell Glioblastoma | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Anaplastic ganglioglioma | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Gliosarcoma | 0 | 0 | 0 | 0 | 0 | 1 | 1
  High Grade Astrocytoma, NOS | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Other, Specify | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Pleomorphic xanthoastrocytoma | 0 | 0 | 0 | 0 | 1 | 0 | 1
WHO 2016 Classification (WHO CNS4) [Count of Participants; unit: Participants] — Patients were graded according to 2016 WHO tumor grading criteria. Grading is based on Histologic + IDH status. HGGs encompass WHO grade III and IV gliomas, including anaplastic astrocytoma (grade 3) and glioblastoma (grade 4).
  Participants
    WHO 2016 Grade 4 | 3 | 3 | 6 | 4 | 62 | 66 | 144
    WHO 2016 Grade 3 | 1 | 0 | 0 | 0 | 18 | 14 | 33
KPS [Count of Participants; unit: Participants] — KPS stands for Karnofsky Performance Status, which is a standard way to measure a patient's ability to perform daily tasks. KPS scores range from 0 to 100, with higher scores indicating a patient is better able to perform daily activities
  Participants
    KPS score 90 | 2 | 1 | 4 | 1 | 39 | 37 | 84
    KPS score 80 | 1 | 1 | 0 | 3 | 22 | 25 | 52
    KPS score 100 | 0 | 0 | 1 | 0 | 19 | 11 | 31
    KPS score 70 | 1 | 1 | 1 | 0 | 0 | 7 | 10

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of BMX-001 Administered in Combination With Standard RT and TMZ in Newly Diagnosed HGG Patients
Description: This was a dose escalation study in which patients were enrolled to receive 1 of 4 doses in dose ascending order. MTD was defined as the dose level that has an estimated DLT rate nearest to 0.25. This is applicable to the Phase 1 part of the study only. Note that an actual MTD was not reached, however a Phase 2 recommended dose was selected based on the dose that was most tolerable to patients.
Time Frame: From the time the subject signs the informed consent form through 30 days after completion of the final BMX-001 treatment (up to approximately 16 weeks)
Population: All patients who received at least 1 dose of BMX-001, regardless of dose level, after enrolling on study.
Measure: Number; unit: mg/Participant
Arm/Group | Phase 1
Number analyzed (Participants) | 17
mg/Participant | NA — MTD was not reached

2. Primary Outcome: Phase 2: Overall Survival, Intent to Treat (ITT) Population
Description: This is applicable for Phase 2 only. It was a secondary objective of Phase 1 and that is reported as a separate outcome measure. Assessment of overall survival. With standard treatment, the median survival of Grade IV patients is expected to be 14.6 months, and the median survival of Grade III is approximately 36 months. Given that we anticipate that approximately 10% of patients to be Grade III, we estimate that the overall median survival with standard treatment to be roughly 16.7 months.
Time Frame: From the time between randomization and death, or the date of last follow-up if the patient remains alive. Per protocol, patients will be followed indefinitely
Population: All enrolled participants enrolled in Phase 2 were included in the analysis. This was not a primary objective of Phase 1.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | ARm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 80 | 80
months | 32.2 [21.8 to NA] — Upper confidence interval was not reached | 27.6 [19.8 to 33.8]
Statistical Analysis 1: Comparison: Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 vs ARm B: Ph 2 Radiation Therapy and TMZ; A 1-tailed logrank test was conducted at the 0.2 level. This test had 90% power to detect a hazard ratio of 0.63 after 84 deaths were observed among the 160 randomized patients; Test type: Superiority; p = 0.135, Log Rank — Study was originally designed with 1 IA after approximately 42 deaths. An unplanned, 2nd IA was conducted to support a BTDR. The study was not terminated early as a result of either IAs. No further IA were conducted until the primary analysis; 89 study participants had passed away at the time of this analysis (41 in the RT/TMZ + BMX-001 arm and 48 in the Radiation Therapy/TMZ arm); Hazard Ratio (HR) = 0.791, 95% CI 1-sided [upper limit 95]

3. Secondary Outcome: Phase 1: Median Overall Survival
Description: Median Overall Survival (OS) is a key clinical outcome measure used to assess the efficacy of BMX-001 in combination with standard radiotherapy (RT) and temozolomide (TMZ) in patients with newly diagnosed high-grade gliomas (HGG). OS is defined as the time from the date of study enrollment to the date of death from any cause. Survival status was assessed at regular follow-up intervals (e.g., every 3 months post-treatment) through medical records, patient contact, and clinical evaluations. The final analysis was conducted after a pre-specified number of events (deaths) have occurred.
  Expected Outcome: Prolonged median OS compared to historical or control data (RT + TMZ alone) would suggest a survival benefit associated with BMX-001.
Time Frame: From the time between enrollment and death, or the date of last follow-up if the patient remains alive.
Population: This analysis includes all participants enrolled. A Kaplan-Meier analysis is not appropriate for very small groups in each dose escalation cohort because the statistical power would be insufficient, leading to unreliable survival estimates. According to the study statistical analysis plan, OS will be assessed for all participants enrolled in Phase 1 as a whole, rather than separately by dose level.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1
Number analyzed (Participants) | 17
Months | 22.2 [11.2 to 24.7]

4. Secondary Outcome: Phase 1: Number of Participants Who Experiences a Dose-limiting Toxicity (DLT).
Description: This is only applicable for the Phase 1 portion of the study. All patients who received at least 1 dose of BMX-001, regardless of dose level, after enrolling on study are included in the analysis.
Time Frame: as for outcome 1
Population: All patients who received at least 1 dose of BMX-001, regardless of dose level, after enrolling on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1
Number analyzed (Participants) | 17
Participants
  BMX-001: 42 mg loading dose / 20 mg biw dose: number analyzed (Participants) | 4
  BMX-001: 42 mg loading dose / 20 mg biw dose | 1
  BMX-001: 28 mg loading dose / 14 mg biw dose: number analyzed (Participants) | 6
  BMX-001: 28 mg loading dose / 14 mg biw dose | 0
  BMX-001: 14 mg loading dose / 7 mg biw dose: number analyzed (Participants) | 3
  BMX-001: 14 mg loading dose / 7 mg biw dose | 0
  BMX-001: 7 mg loading dose / 3.5 mg biw dose: number analyzed (Participants) | 4
  BMX-001: 7 mg loading dose / 3.5 mg biw dose | 0

5. Secondary Outcome: Phase 1: Examine the Impact on Cognition of BMX-001 in Combination With Standard RT and TMZ in Treatment of Newly Diagnosed HGG Patients Via the Adjusted Change T Score Achieved on the Controlled Oral Word Association Test (COWAT).
Description: The Controlled Oral Word Association Test (COWAT) measures verbal fluency which reflects executive functioning, processing speed, mental flexibility, and language output.
  The raw score is then adjusted for age, education, and normative data to allow meaningful comparisons across individuals. The standardized score (T-score) is calculated using normative reference tables.
  Higher Scores = Better Cognitive Function, lower scores = cognitive impairment. T score range is 0-100.
  A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean performance with a standard deviation of 10.
  T-scores below 40 suggest clinically significant cognitive decline. Scores range from < 30 (significantly below average), to 30-39 (below average), 40-59 (average), and greater than or equal to 60 is above average.
  Stable or improved COWAT scores over time would suggest that adding BMX-001 may help preserve cognitive function.
Time Frame: From the time the subject signs the informed consent form through 6 months after completion of the final BMX-001 treatment (up to approximately 40 weeks)
Population: Only 6 out of 17 eligible participants completed COWAT assessments at the time this objective was measured 24 weeks after the end of standard of care Radiotherapy + Temozolomide.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 1
Number analyzed (Participants) | 6
T-score
  BMX-001: 7 mg loading dose / 3.5 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 7 mg loading dose / 3.5 mg biw dose | 4 (NA) — Sample size is 1
  BMX-001: 14 mg loading dose / 7 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 14 mg loading dose / 7 mg biw dose | -3 (NA) — Sample size is 1
  BMX-001: 28 mg loading dose / 14 mg biw dose: number analyzed (Participants) | 3
  BMX-001: 28 mg loading dose / 14 mg biw dose | 2 (9.6)
  BMX-001: 42 mg loading dose / 20 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 42 mg loading dose / 20 mg biw dose | 22 (NA) — Sample size is 1

6. Secondary Outcome: Phase 1: Examine the Impact on Cognition of BMX-001 in Combination With Standard RT and TMZ in Treatment of Newly Diagnosed HGG Patients Via the Normalized Score Achieved on the Trails Making Test (TMT): Part A
Description: Part A of the Trails Making Test (TMT) measures visual attention and processing speed by requiring the patient to connect numbers sequentially (1 → 2 → 3, etc.) as quickly as possible. This is a widely used neuropsychological test that measures visual attention, processing speed, and psychomotor function.
  Raw scores are measured in seconds (time to complete the task), but T-scores are derived by converting time-based results into a normed distribution accounting for age and education.
  Mean (SD) change in cognitive assessment in T-Scores is reported and the range is 0-100.
  T score interpretation and range is < 30 (significantly impaired), 30-39 (mildly impaired), 40-59 (Average), >/= 60 (Above average). A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean performance with a standard deviation of 10.
  Higher scores = better performance.
Time Frame: as for outcome 5
Population: Only 6 out of 17 eligible participants completed Trail Making Test (TMT): Part A assessments at the time this objective was measured 24 weeks after the end of standard of care Radiotherapy + Temozolomide.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Phase 1
Number analyzed (Participants) | 6
T-Score
  BMX-001: 7 mg loading dose / 3.5 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 7 mg loading dose / 3.5 mg biw dose | -0.4 (NA) — Sample size is 1
  BMX-001: 14 mg loading dose / 7 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 14 mg loading dose / 7 mg biw dose | 5.1 (NA) — Sample size is 1
  BMX-001: 28 mg loading dose / 14 mg biw dose: number analyzed (Participants) | 3
  BMX-001: 28 mg loading dose / 14 mg biw dose | 0.9 (0.4)
  BMX-001: 42 mg loading dose / 20 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 42 mg loading dose / 20 mg biw dose | 3.1 (NA) — Sample size is 1

7. Secondary Outcome: Phase 1: Examine the Impact on Cognition of BMX-001 in Combination With Standard RT and TMZ in Treatment of Newly Diagnosed HGG Patients Via the Normalized Score Achieved on the Trail Making Test (TMT): Part B
Description: The Trails Making Test (TMT) Part B is a widely used neuropsychological test that measures set-shifting ability, processing speed, and working memory. While Part A focuses on speed, visual scanning, and attention.
  Prolonged completion time or an increase in errors compared to baseline or age-adjusted norms would indicate cognitive decline.
  Raw scores are measured in seconds (time to complete the task), but T-scores are derived by converting time-based results into a normed distribution accounting for age and education.
  Mean (SD) change in T score is reported, range is 0-100. T score interpretation and range is < 30 (significantly impaired), 30-39 (mildly impaired), 40-59 (Average), >/= 60 (Above average). A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean performance with a standard deviation of 10.
  Higher scores = better performance.
Time Frame: as for outcome 5
Population: Only 6 out of 17 eligible participants completed Trail Making Test (TMT): Part B assessments at the time this objective was measured 24 weeks after the end of standard of care Radiotherapy + Temozolomide.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 1
Number analyzed (Participants) | 6
T-score
  BMX-001: 7 mg loading dose / 3.5 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 7 mg loading dose / 3.5 mg biw dose | 0.3 (NA) — Sample size is 1
  BMX-001: 14 mg loading dose / 7 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 14 mg loading dose / 7 mg biw dose | 7.1 (NA) — Sample size is 1
  BMX-001: 28 mg loading dose / 14 mg biw dose: number analyzed (Participants) | 3
  BMX-001: 28 mg loading dose / 14 mg biw dose | -0.3 (1)
  BMX-001: 42 mg loading dose / 20 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 42 mg loading dose / 20 mg biw dose | 1 (NA) — Sample size is 1

8. Secondary Outcome: Phase 1: Examine the Impact on Cognition of BMX-001 in Combination With Standard RT and TMZ in Treatment of Newly Diagnosed HGG Patients Via the Normalized Total Recall Change T-score Achieved on the Hopkins Verbal Learning Test- Revised (HVLT-R)
Description: Hopkins Verbal Learning Test- Revised (HVLT-R) is a standardized neuropsychological assessment that measures verbal learning and memory, including total (immediate recall). Total Recall T-score is derived from the sum of correctly recalled words across three learning trials and is normalized based on age-adjusted normative data. This provides insight into immediate verbal memory performance and learning ability.
  Total Recall (Immediate Memory & Learning) is Sum of correctly recalled words across three learning trials and is a measurement of immediate recall capacity and learning efficiency.
  Raw score range is 0-36, T score range is 0-100. T scores >/= 60 are above average and T scores < 40 are below average. A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean with a standard deviation of 10
Time Frame: as for outcome 5
Population: Only 6 out of 17 eligible participants completed HVLT-R assessments at the time this objective was measured 24 weeks after the end of standard of care Radiotherapy + Temozolomide.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Phase 1
Number analyzed (Participants) | 6
T-Score
  BMX-001: 7 mg loading dose / 3.5 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 7 mg loading dose / 3.5 mg biw dose | 17 (NA) — Sample size is 1
  BMX-001: 14 mg loading dose / 7 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 14 mg loading dose / 7 mg biw dose | -5 (NA) — Sample size is 1
  BMX-001: 28 mg loading dose / 14 mg biw dose | -1 (11.4)
  BMX-001: 42 mg loading dose / 20 mg biw dose: number analyzed (Participants) | 1
  BMX-001: 42 mg loading dose / 20 mg biw dose | 19 (NA) — Sample size is 1

9. Secondary Outcome: Phase 2: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: To assess the safety and tolerability of standard RT and TMZ in combination with BMX-001 compared to standard RT and TMZ alone in newly diagnosed HGG patients. The phase 2 portion of this study has two adverse event endpoints:
  1. The proportion of patients who experience any grade 3 or 4 adverse event during radiation and temozolomide treatment, and
  2. The proportion of patients who experience a grade 3 or 4 adverse event that is definitely, possibly, or probably related to BMX-001 treatment during this same period.
  This outcome measure does not apply to the Phase 1 portion of the study, as it was not designated as an outcome for Phase 1 but was specified only for Phase 2.
Time Frame: Adverse events occurring from baseline through 30 days post completion of treatment (approximately 12 weeks total).
Population: This analysis focuses on the proportion of patients who experience any grade 3 or 4 adverse event during radiation and temozolomide treatment.
  This outcome measure does not apply to the Phase 1 portion of the study, as it was not designated as an outcome for Phase 1 but was specified only for Phase 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 80 | 80
Participants | 17 | 13

10. Secondary Outcome: Phase 2: Incidence of Treatment-Emergent Adverse Events Related to BMX-001
Description: To assess the safety and tolerability of standard RT and TMZ in combination with BMX-001 compared to standard RT and TMZ alone in newly diagnosed HGG patients.
  This outcome is measured to test the proportion of patients who experience a grade 3 or 4 adverse event that is definitely, possibly, or probably related to BMX-001 treatment during this same period.
  This outcome measure does not apply to the Phase 1 portion of the study, as it was not designated as an outcome for Phase 1 but was specified only for Phase 2. It also only applies to Arm A in the study as Arm B did not receive the study drug.
Time Frame: Adverse events occurring from baseline through 30 days post completion of treatment (approximately 12 weeks total).
Population: This outcome measure does not apply to the Phase 1 portion of the study, as it was not designated as an outcome for Phase 1 but was specified only for Phase 2.
  This analysis focuses on the proportion of patients who experience a grade 3 or 4 adverse event that is definitely, possibly, or probably related to BMX-001 treatment during this same period. Data is only presented for Arm A, the BMX-001 treatment group, as subjects in Arm B did not receive BMX-001.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001
Number analyzed (Participants) | 80
Participants | 5

11. Secondary Outcome: Phase 2: Protection/Improvement of Cognition Using Hopkins Verbal Learning-Revised
Description: Hopkins Verbal Learning Test- Revised (HVLT-R) is a standardized neuropsychological test that measures verbal learning and memory, including total (immediate recall), delayed recall, and recognition discrimination. It is scored using a T-score which are calculated based on raw scores (e.g., number of words recalled) and standardized using normative data adjusted for age, education, and sometimes sex. T-score range is 0-100. T-scores >/= 60 are above average and T scores < 40 are below average. Higher scores are better. Total recall interpretation - T ≥ 60: above average; T < 40: below average. Delayed recall - T < 30 may suggest memory consolidation issues, and recognition discrimination - T < 30 may indicate impaired recognition memory. A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean performance with a standard deviation of 10.
  Mean (SD) change in cognitive assessment is reported.
Time Frame: Baseline and Week 24
Population: Only patients that had both a baseline + follow up tests completed could be included in the analysis
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 80 | 80
T-Score
  HVLT-R Delayed Recall T Score: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radrx Compltion: number analyzed (Participants) | 29 | 14
  HVLT-R Delayed Recall T Score: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radrx Compltion | 0.45 (13.18) | -4.07 (8.61)
  HVLT-R Recognition Index T Score: Mean Changes from Bseline at Wk 24 (+/-4 Wks) Post-radrx Compltion: number analyzed (Participants) | 29 | 14
  HVLT-R Recognition Index T Score: Mean Changes from Bseline at Wk 24 (+/-4 Wks) Post-radrx Compltion | -2.14 (13.81) | 2.79 (11.77)
  HVLT-R Retention T Score: Mean Changes from Baseline at Week 24 (+/-4 Weeks) Post-radrx Completion: number analyzed (Participants) | 29 | 14
  HVLT-R Retention T Score: Mean Changes from Baseline at Week 24 (+/-4 Weeks) Post-radrx Completion | 1.79 (15.49) | -2.29 (16.06)
  HVLT-R Total Recall T Score: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radrx Completion: number analyzed (Participants) | 29 | 14
  HVLT-R Total Recall T Score: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radrx Completion | 2 (9.82) | 0.07 (13.85)

12. Secondary Outcome: Phase 2: Protection/Improvement of Cognition Via the Controlled Oral Word Association Test (COWAT)
Description: This Controlled Oral Word Association Test (COWAT) measure verbal fluency which reflects executive functioning, processing speed, mental flexibility, and language output.
  The raw score is adjusted for age, education, and normative data to allow meaningful comparisons across individuals. The standardized score (T-score) is calculated using normative reference tables.
  Higher Scores = Better Cognitive Function, lower scores = cognitive impairment. T-score range is 0-100 A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean performance with a standard deviation of 10.
  T-scores below 40 suggest clinically significant cognitive decline. Scores range from < 30 (significantly below average), to 30-39 (below average), 40-59 (average), and greater than or equal to 60 is above average.
  Stable or improved COWAT scores over time would suggest that adding BMX-001 may help preserve cognition.
Time Frame: Baseline and Week 24
Population: Only patients that had both a baseline + follow up tests completed could be included in the analysis
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 27 | 13
T-Score | 4.19 (14.65) | 5.23 (11.2)

13. Secondary Outcome: Phase 2: Protection/Improvement of Cognition - Trails Making Test A and B
Description: Phase 1 is reported separately. Neurocognitive testing was done and reported here for the Trails Test A and B Part A: Visual attention and processing speed Part B: Executive functioning, task switching, and divided attention. Part A testing time is typically 20-90 sec, and Part B time is typically 40-180 sec.
  Raw scores are measured in seconds (time to complete the task), but T-scores are derived by converting time-based results into a normed distribution accounting for age and education.
  Mean (SD) change in cognitive assessment in T-Scores is reported T score interpretation and range is < 30 (significantly impaired), 30-39 (mildly impaired), 40-59 (Average), >/60 (above average) A T-score of 50 represents the mean performance in the normative population, this means a score of 50 indicates the population mean performance with a standard deviation of 10.
  Lower times = better
Time Frame: Baseline and Week 24 Baseline and Week 24 Baseline and Week 24
Population: Only patients that had both a baseline + follow up tests completed could be included in the analysis
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 80 | 80
T Score
  Trail A Completion Time: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radiation Completion: number analyzed (Participants) | 28 | 14
  Trail A Completion Time: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radiation Completion | -0.24 (2.08) | 2.37 (6.45)
  Trail B Completion Time: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radiation Completion: number analyzed (Participants) | 28 | 14
  Trail B Completion Time: Mean Changes from Baseline at Week 24 (+/-4 Wks) Post-radiation Completion | .19 (1.33) | 2.29 (4.46)

14. Secondary Outcome: Phase 2: Protection of Bone Marrow Against Chemotherapy-Induced Thrombocytopenia
Description: This was not a secondary outcome in Phase 1 and therefore only applies to Phase 2. The proportion of patients who experience grade 3 or 4 thrombocytopenia during concurrent temozolomide and radiation will be recorded within each treatment group. The proportion of patients who experience a platelet count less than 100K during concurrent temozolomide and radiation will also be recorded within each treatment group. For both endpoints described above, a chi-square or Fisher's exact test was conducted to compare the prevalence of such thrombocytopenia observed in patients with and without BMX-001.
Time Frame: Approximately 12 weeks (from Baseline to 30 days post completion of treatment)
Population: For this endpoint to have relevance, a patient must have received some treatment with temozolomide and radiation in either Arm A or B. Analyses suggest that 78 patients in Arm A and 71 patients in Arm B received at least some form of protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 78 | 71
Participants | 1 | 2
Statistical Analysis 1: Comparison: Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 vs Arm B: Ph 2 Radiation Therapy and TMZ; With 78 and 71 patients in Arms A and B, respectively, there was 80% power with a one-tailed chi-square test (α=0.05) to detect a reduction in grade 3 or 4 thrombocytopenia from 15% in Arm B (without BMX-001) to 3.7% in Arm A (with BMX-001). Given the small number of patients that experienced low platelet counts or thrombocytopenia, a one-tailed Fisher's exact test was performed instead; Test type: Superiority; p = 0.465, Fisher Exact; Odds Ratio (OR) = 0.45

15. Secondary Outcome: Phase 1 and Phase 2: Progression-free Survival (PFS)
Description: The primary analysis of PFS will consider all patients, and consider them in their assigned treatment arm regardless of compliance. This approach to analysis is consistent with an intent-to-treat analysis approach. Progression-Free Survival (PFS) is defined as the time from randomization (Phase 2) or study enrollment (Phase 1) to the first occurrence of either disease progression (as determined by standardized radiographic criteria, the RANO [Response Assessment in Neuro-Oncology] criteria) or death from any cause, whichever occurs first. Patients who have not experienced progression or death at the time of analysis will be censored at their last known follow-up date. PFS will be estimated using the Kaplan-Meier method, providing median PFS and corresponding 95% confidence intervals (CI).
Time Frame: up to 5 years
Population: All patients enrolled in each specific arm
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Phase 1: All subjects enrolled in the Phase 1 dose escalation portion of the study.
Arm/Group | Phase 1 | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 17 | 80 | 80
months | 7.1 [3.9 to 11.4] | 11.9 [8.4 to 28.4] | 14.7 [9.6 to 28.5]
Statistical Analysis 1: Comparison: Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 vs Arm B: Ph 2 Radiation Therapy and TMZ; A 1-tailed logrank test was conducted at the 0.2 level; Test type: Superiority; p = 0.911, Log Rank; Hazard Ratio (HR) = 0.978

16. Secondary Outcome: Phase 1 and 2: Complete or Partial Radiographic Response to Tumor
Description: The guidelines and criteria for radiographic response will be based on the updated RANO criteria for newly diagnosed GBM. MRI brain with and without contrast will be obtained at enrollment, 2-4 weeks after standard RT and TMZ, and every 8 weeks during adjuvant TMZ. Since this is a study in newly diagnosed patients with HGG, the baseline imaging will be designated as the imaging obtained 2 to 4 weeks after the completion of standard RT and TMZ. At each time point, based on RANO criteria, the subject response will be characterized as Complete Response, Partial Response, Progressive Disease, Stable Disease, or Not Evaluable.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Phase 1: Dose escalation cohort
Arm/Group | Phase 1 | Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 | Arm B: Ph 2 Radiation Therapy and TMZ
Number analyzed (Participants) | 17 | 80 | 80
proportion of participants | 0 [0 to 0] | 0.1125 [0.0528 to 0.2028] | 0.0625 [0.0206 to 0.1399]
Statistical Analysis 1: Comparison: Arm A: Ph 2 Radiation Therapy, TMZ and BMX-001 vs Arm B: Ph 2 Radiation Therapy and TMZ; Test type: Superiority; p = 0.401, Chi-squared, Corrected; A continuity adjusted Chi-Squared test was performed

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events relating to investigational treatment for 12 weeks, patients were monitored for vital status for up to 5 years
Groups:
- Phase 1: BMX-001: 7 mg Loading Dose / 3.5 mg Biw Dose: The dose escalation study. Patients will receive standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 7 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks
- Phase 1: BMX-001: 14 mg Loading Dose / 7 mg Biw Dose: The dose escalation study. Patients will receive standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 14 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks
- Phase 1: BMX-001: 28 mg Loading Dose / 14 mg Biw Dose: The dose escalation study. Patients will receive standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks
- Phase 1: BMX-001: 42 mg Loading Dose / 20 mg Biw Dose: The dose escalation study. Patients will receive standard of care radiation therapy plus temozolomide (TMZ). BMX-001 was given by subcutaneous injection with a loading dose of42 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks
- Arm A: Radiation Therapy, TMZ and BMX-001: Patients will receive standard of care radiation therapy plus temozolomide (TMZ). BMX-001 will be given by subcutaneous injection with a loading dose of 28 mg/subject given within 4 days prior to initiation of radiation therapy and followed by biweekly maintenance doses at half the loading dose for a total of 8 weeks. A total of 80 subjects will receive BMX-001 in this phase.
  BMX-001: BMX-001 consists of a porphyrin ring with pyridyl groups attached at each of the four methane bridge carbons. The nitrogen in the pyridyl ring is at the 2 position and has a side chain consisting of six carbons with an ether linkage. A manganese atom is chelated into the porphyrin ring and is the active center of the molecule. This molecule is an enzymatic scavenger of free radical species operating at close to diffusion-limited rates.
  Radiation Therapy: RT will be delivered in daily fractions of 1.8-2 Gy given 5 days a week for 6 weeks for a total of 59.4-60 Gy.
  Temozolomide: Initially, temozolomide (TMZ) will be dosed at 75 mg/m2 orally daily for 42 days. Two weeks after the completion of chemoradiation, patients will transition to adjuvant chemotherapy with TMZ dosed at 150-200 mg/m2 orally for 5 days of a 28-day cycle for a total of 12 cycles.
- Arm B: Radiation Therapy and TMZ: In this arm, one-half of the study subjects will not receive BMX-001 but will undergo all components of standard therapy (radiation therapy plus temozolomide [TMZ]). A total of 80 subjects will be in this study arm.
  Radiation Therapy: RT will be delivered in daily fractions of 1.8-2 Gy given 5 days a week for 6 weeks for a total of 59.4-60 Gy.
  Temozolomide: Initially, temozolomide (TMZ) will be dosed at 75 mg/m2 orally daily for 42 days. Two weeks after the completion of chemoradiation, patients will transition to adjuvant chemotherapy with TMZ dosed at 150-200 mg/m2 orally for 5 days of a 28-day cycle for a total of 12 cycles.
Arm/Group | Phase 1: BMX-001: 7 mg Loading Dose / 3.5 mg Biw Dose | Phase 1: BMX-001: 14 mg Loading Dose / 7 mg Biw Dose | Phase 1: BMX-001: 28 mg Loading Dose / 14 mg Biw Dose | Phase 1: BMX-001: 42 mg Loading Dose / 20 mg Biw Dose | Arm A: Radiation Therapy, TMZ and BMX-001 | Arm B: Radiation Therapy and TMZ
All-Cause Mortality (participants affected / at risk) | 3/4 | 3/3 | 6/6 | 4/4 | 41/80 | 48/80
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/3 | 0/6 | 2/4 | 11/80 | 10/80
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 6/6 | 4/4 | 77/80 | 70/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: BMX-001: 7 mg Loading Dose / 3.5 mg Biw Dose (N=4) | Phase 1: BMX-001: 14 mg Loading Dose / 7 mg Biw Dose (N=3) | Phase 1: BMX-001: 28 mg Loading Dose / 14 mg Biw Dose (N=6) | Phase 1: BMX-001: 42 mg Loading Dose / 20 mg Biw Dose (N=4) | Arm A: Radiation Therapy, TMZ and BMX-001 (N=80) | Arm B: Radiation Therapy and TMZ (N=80)
Dyspnoea (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 4
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 3
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Muscular weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: BMX-001: 7 mg Loading Dose / 3.5 mg Biw Dose (N=4) | Phase 1: BMX-001: 14 mg Loading Dose / 7 mg Biw Dose (N=3) | Phase 1: BMX-001: 28 mg Loading Dose / 14 mg Biw Dose (N=6) | Phase 1: BMX-001: 42 mg Loading Dose / 20 mg Biw Dose (N=4) | Arm A: Radiation Therapy, TMZ and BMX-001 (N=80) | Arm B: Radiation Therapy and TMZ (N=80)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 5 | 2 | 22 | 14
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0 | 0 | 2 | 17 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 8 | 0
Auditory disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 1 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 3
Labyrinthitis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Middle ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Otitis externa (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0
Accommodation disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 0
Pupillary disorder (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Quadrantanopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 4
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 2 | 1 | 30 | 30
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 10 | 10
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 4 | 3
Hiccups (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 1 | 4 | 1 | 45 | 27
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 11 | 9
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 2 | 3 | 0
Fatigue (General disorders) | 0 | 2 | 5 | 2 | 49 | 41
Incision site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site hypersensitivity (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site papule (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site urticaria (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 4 | 4
Pain (General disorders) | 0 | 0 | 3 | 0 | 7 | 3
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 16 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Helicobacter gastritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Incision site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 5 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 3 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 4 | 5
Injection site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Injection site paraesthesia (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Injection site pruritus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Injection site reaction (Injury, poisoning and procedural complications) | 2 | 3 | 2 | 0 | 64 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 2 | 14 | 9
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 2 | 11 | 11
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Blood bilirubin (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1 | 4 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 1 | 0 | 3 | 5
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 4
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT interval (Investigations) | 0 | 0 | 0 | 0 | 3 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Granulocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 6 | 2
Granulocyte percentage (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Haematocrit decreased (Investigations) | 0 | 0 | 0 | 0 | 3 | 4
Haematocrit increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Lipase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 4 | 2 | 24 | 21
Lymphocyte percentage decreased (Investigations) | 0 | 0 | 0 | 0 | 7 | 6
Mean cell haemoglobin concentration (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 2 | 1 | 6 | 4
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 0
Neutrophil percentage increased (Investigations) | 0 | 0 | 0 | 0 | 4 | 1
Platelet count decreased (Investigations) | 2 | 1 | 5 | 2 | 19 | 14
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 7 | 4
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 3
White blood cell count decreased (Investigations) | 1 | 0 | 3 | 2 | 7 | 6
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 8 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 13 | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 2 | 12 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 5
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 4 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 1 | 5 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1 | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 2 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 7 | 9
Oedema (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 5 | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 3
Chills (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 3
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 4
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 3 | 1 | 10 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0 | 8 | 8
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gait disturbance (Nervous system disorders) | 0 | 0 | 1 | 0 | 4 | 3
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 2 | 0 | 18 | 20
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 5 | 0
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 11 | 5
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 2 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 3 | 7
Pyramidal tract syndrome (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 2
Seizure (Nervous system disorders) | 0 | 1 | 1 | 2 | 9 | 7
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Subdural hygroma (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Nervous system disorders) | 0 | 0 | 2 | 1 | 4 | 3
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 6
Visual field defect (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 9 | 7
Aphasia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 5 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 6 | 6
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2
Dysarthria (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 2
Hypersomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 6 | 8
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 4 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 2 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2 | 0
Anosmia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 4 | 9
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 5 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 5 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 0 | 33 | 26
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0 | 4 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 2
Injection site discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 21 | 3
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Radiation skin injury (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 5 | 5
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin sensitisation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 5 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Constipation prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 6 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 8 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 3 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Barotitis media (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 2
Nystagmus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Brain oedema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Monocyte percentage increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Neurological examination abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Autonomic nervous system imbalance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Eyelid ptosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Intention tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pseudomeningocele (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Restlessness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vertigo (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Disturbance in attention (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Memory impairment (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 8
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2
Laceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 9
Incision site haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0
Fecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fecal Urgency (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
GASSY, ABDOMINAL PAIN AND FEELING FLUSHED (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
PIMPLE LIKE SORE (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Shingles (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
EMOTIONAL LABILITY (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash acnneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Cold (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Dry sinuses (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flu like symptoms (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Head cold (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT02655601/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT02655601/SAP_001.pdf
  • Informed Consent Form (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/01/NCT02655601/ICF_002.pdf